CLINICAL TRIAL: NCT07354386
Title: Researcher-blinded Randomized Controlled Trial of the Effects of Dried Whole Fruits on Glucose and Lipid Levels in Prediabetic and Type 2 Diabetic Individuals
Brief Title: Effects of Dried Whole Fruits on Metabolism in Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS26882 (B2025:027)
Record Dates: First submitted 2026-01-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes; Type 2 Diabetes
Keywords: Saskatoon berry; Dried apple; Fasting plasma glucose; Lipids; Insulin resistance; Inflammatory markers; Gut microbiota
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze dried whole Saskatoon berry (Experimental): Freeze dried whole Saskatoon berry 40 g/day for 12 weeks
  Interventions: Dietary Supplement: Freeze dried whole Saskatoon berry
- Freeze dried apple slize bulk (Placebo Comparator): Freeze dried apple slice bulk in the same carbohydrate amount as in 40 g of Saskatoon berry per day for 12 weeks
  Interventions: Dietary Supplement: Freeze dried apple slice bulk

INTERVENTIONS:
Dietary Supplement: Freeze dried whole Saskatoon berry — Freeze dried whole Saskatoon berry 40 g/day for 12 weeks
  Arms: Freeze dried whole Saskatoon berry
Dietary Supplement: Freeze dried apple slice bulk — Freeze dried apple slice bulk in same carbohydrate amount as 40 g Saskatoon berry per day for 12 weeks
  Arms: Freeze dried apple slize bulk

SUMMARY:
Diabetes becomes epidemic in worldwide countries. Diabetes Canada indicated that 30% of adults in Manitoba are diabetes or prediabetes. Nine out of ten diabetic patients are type 2 diabetes (T2D). T2D is characterized by insulin resistance and obesity. Uncontrolled diabetes leads to serious consequences including heart attack, stroke, chronic renal failure, liver failure, blindness and low limb amputation. Most of hypoglycemic medications have certain side effects. Natural foods or nutraceuticals with hypoglycemic potential are expected to provide a safer management for diabetic patients. Saskatoon berry is a popular fruit in Canadian Prairie and Northern states in USA. Previous studies in the investigator's group demonstrated Saskatoon berry (SB) powder attenuated hyperglycemia, hyperlipidemia, insulin resistance, inflammation, liver steatosis and gut dysbiosis in diet-induced insulin resistant mice, a model for T2D. The findings of the glucose and lipid lowering or liver protective effects of SB powder have been supported by another group in Australia in high fat fed rats. Preliminary studies by the investigators in 20 healthy subjects demonstrated that dried whole SB (40 g/day for 10 weeks) significantly reduced fasting plasma glucose, total and LDL-cholesterol, systolic blood pressure, and increased plasma glucagon-like peptide compared to baseline, which was associated with increased intake of total fiber and decreased intake of saturated fat. The changes in metabolic and vascular variables significantly correlated with the alterations in gut microbiota The combination of findings suggest that SB is good candidate of prebiotic functional food as a supplemental remedy for reducing the risk for metabolic syndrome and preventing or managing T2D. The effect of Saskatoon berry and its products on metabolic disorders have not been studied in diabetic subjects. The investigators propose to examine the effects of oral administration of freeze-dried whole SB on glucose metabolism, insulin resistance and gut microbiota in untreated prediabetes and new type 2 diabetic patients compared to a control dried fruit in a randomized controlled trial.

DETAILED DESCRIPTION:
Subject recruitment: Untreated prediabetes or new type 2 diabetic (T2D) patients (males and females, 18-74 years of age) and willing to sign an informed consent will be recruited from community clinics in Winnipeg, Endocrine or Hepatologic Clinics in University of Manitoba and Rossmere Medical Centre in Winnipeg by posters. Exclusion criteria include: 1) candidates have a history of myocardial infarction, stroke or chronic kidney disease; 2) participants treated with hypoglycemic, anti-hypertensives, lipid lowering medications or antibiotics within a month. Candidates will be invited to read and voluntarily sign an informed consent approved by Research Ethics Board in University of Manitoba. Recruitment goal: n = 92 (80 + 15% expected drop-off).

Randomization: Eligible participant will be enrolled and randomization into two groups through a web randomization tool. Randomized ID will be obtained for each participant used in files or labels on packages of dried fruits.

Dietary supplements: Freeze dried Saskatoon berry (SB) have been obtained from Prairie Berries Inc. The berries were freshly frozen and no supplementation was added to the dried berry. The product has been processed by certified facilities and the batch of dried berry has passed pathogen analysis. Control dietary supplement will be dried apple slice bulk without supplementation (Vancouver Freeze Dry, Langley, BC). Two types of dietary supplements will be weighed and packed: 1) 40 g of dried whole SB/bag; 2) dried apple slice bulk in a weight containing carbohydrate equivalent to 40 g of SB/bag). Non-transparent bags labeled only with randomization ID will be used for the package of the fruits.

Duration of the dietary regimen: 12 weeks.

Scheduled visits:

Visit 1: Consent and enrollment. A questionnaire for domestic questionnaire including dietary intake and physical activity will be filled. Measurements of body weight, height and blood pressure will be taken during the visit.

Visit 2 (<1 week from the visit 1 and before the start of berry administration): Blood withdrawal at Health Sciences Center (HSC) in Winnipeg after an overnight fasting. Fasting plasma glucose, insulin, HbA1C, lipid profile, liver enzymes (alanine transaminase or ALT, aspartate transaminase or AST), apoB, apoA-I, and creatinine will be analyzed in Clinical Chemistry in HSC. An extra 3 ml of blood withdraw in serum tube. The serum will be temporarily stored in Clinical Chemistry for measuring insulin, GLP-1 and high-sensitive C-reactive protein (hs-CRP) by Investigator's group.

Visit 3 (at 6 weeks after the start of administration of Saskatoon berry): Participants will be asked to provide feedback on general well-being and the intake of Saskatoon berry. Body weight, blood pressure and heart rate will be measured and recorded.

Visit 4 (at 12 weeks after the start of the dietary regimen): Participants will be asked to collect stool sample with the collection kit within 1 week before the visit and bring it to the visit. They will also be asked to have an overnight fasting the night before visit. Blood samples will be collected for biochemical analyses as descried in Visit 2. Same amount blood will be collected for serum temporarily stored for the analysis of GLP-1 and hs-CRP. During the visit, body weight, blood pressure and heart rate of participants will be taken. Questionnaires on participants' dietary intake, physical activity and feedback to the study will be completed. Homeostatic model assessment-insulin resistance or homeostatic model assessment for insulin resistance (HOMA-IR) will be calculated based on fasting plasma glucose and insulin. Stool samples will be aliquoted and stored under -80°C before shipment to analysis in Integrate Microbiome Resource at Dalhousie University.

Data collection and analysis: Biochemical, physical exam, questionnaires, surveys, results from gut microbiota and SCFAs will be collected and inputted to password protected computers of PI and Project Coordinator with only ID but not names or other identifiable information. Data will be analyzed using standards statistical software and tools.

Expected outcomes Primary outcome: Fasting plasma glucose at the end of 12 weeks of SB intake compared to baseline.

Secondary outcomes: HBA1c, fasting serum total cholesterol, LDL-cholesterol, triglyceride, insulin resistance, GLP-1, AST, ALT, CAP (fibroscan), creatinine, hs-CRP, SBP and DBP at the end of 12 weeks of SB intake versus baseline.

ELIGIBILITY:
Inclusion Criteria:

* Untreated pre-diabetes with or without fatty liver disease
* Untreated type 2 diabetes with or without fatty liver disease
* Males and females (18-74 years)
* Signed informed consent

Exclusion Criteria:

* Treated with hypoglycemic, hypolipidemic, anti-hypertensive or antibiotics within 1 month
* Acute myocardial infarction, stroke, heart failure, chronic kidney disease, cirrhosis, metastatic cancers
* Currently pregnancy or nursing
* Allergy to fruits

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG) | 12 weeks
  FPG (mM/L, normal range 3.6-6.1 mM/L) will be measured chemically at baseline and end of the intervention

SECONDARY OUTCOMES:
Hemaglobin A1C (HbA1c) | 12 weeks
  Fasting blood HbA1c (%, normal range 4.0-6.0%) will be measured chemically at the baseline and the end of the intervention
Total serum choleserol (TC) | 12 weeks
  Fasting TC (mM/L. normal for adults <5.2 mM/) will be measured chemically at the baseline and the end of the intervention.
Low density lipoprotein-cholesterol (LDL-c) | 12 weeks
  Fasting LDL-c (mM/L, normal <2 mM/L) will be measured chemically at the baseline and the end of the intervention.
Triglycerides (TAG) | 12 weeks
  Fasting serum TAG (mM/L, normal <1.7 mM/L) will be measured chemically at the baseline and the end of the intervention.
High density lipoprotein-cholesterol (HDL-c) | 12 weeks
  Fasting serum HDL-c (mM/L, normal >1.0 mM/L) will be measured chemically at the baseline and the end of the intervention.
Apoprotein B (apoB) | 12 weeks
  Fasting serum apoB (g/L, normal <1.2 g/L) will be measured chemically at the baseline and the end of the intervention.
Apoprotein A-I (apoA-I) | 12 weeks
  Fasting serum apoA-I (gL, normal male adults >1.07 g/L. normal female >1.22 g/L) will be measured chemically at the baseline and the end of the intervention.
Insulin | 12 weeks
  Fasting serum insulin (pmol/L, normal <140 pmol/L) will be measured chemically at the baseline and the end of the intervention.
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | 12 weeks
  HOMA-IR is an adjusted ratio based on FPG and fasting insulin in simultaneously collected blood samples (normal <1.9) and it will be calculated for samples collected at the baseline and the end of the intervention.
Glucagon-like peptide-1 (GLP-1) | 12 weeks
  Fasting serum GLP-1 (pmol/L, normal 015 pmol/L) will be measured using MSD V-Plex GLP-1 active kit at the baseline and the end of the intervention.
High-sensitive C-reative protein (hs-CRP) | 12 weeks
  Fasting plasma hs-CRP (mg/L, normal <10 mg/L) will be measured using ELISA kit at the baseline and the end of the intervention.
Aspartate transaminase (AST) | 12 weeks
  Serum AST (U/L, normal range 10-32 U/L) will be measured chemically at the baseline and the end of the intervention.
Alanine transaminase (ALT) | 12 weeks
  Serum ALT (U/L, normal range: male < 30 U/L, female < 25 U/L) will be measured chemically at the baseline and the end of the intervention.
Conditioned Attenuation Paramer (CAP) from fibroscan | <12 months
  CAP (dB/m, normal range <238 dB/m) will be assessed <3 months after the end of the dietary intervention compared to that measured <6 months before the start of the intervention in Hepatology Clinic.
Systolic blood pressure (SBP) | 12 weeks
  SBP (mmHg, normal <130 mmHg) will be measured at sitting position after >5 min of rest at baseline and at the end of intervention
Diastolic blood pressure (DBP) | 12 weeks
  DBP (mmHg, normal range 60-80 mmHg) will be measured at sitting position after >5 min of rest at baseline and at the end of intervention
Body weights | 12 weeks
  Body weights (kg) will be measured will be measured at baseline and at the end of intervention. Body weight will be used to calculate body mass index (BMI) using height of the same participant. The normal range of BMI is 18.5-24.9 kg/M2.
Gut microbiome | 12 weeks
  Gut microbiome will be analysed in fecal samples collected at baseline and at the end of intervention at Dalhousie University to determine bacterial composition, abundance and relationship with metabolism. The normal range of human gut microbiome currently does not available.
Fecal short chain fatty acids (SCFA) | 12 weeks
  Fecal SCFA will be analysed in fecal samples collected at baseline and at the end of intervention by Microbiome Insight Inc. to determine fecal SCFA composition, abundances and relationship with metabolism. The normal range of human fecal SCFA currently does not available.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Participants' privacy and confidential information would not be disclosed.

REFERENCES:
- [Background] du Preez R, Wanyonyi S, Mouatt P, Panchal SK, Brown L. Saskatoon Berry Amelanchier alnifolia Regulates Glucose Metabolism and Improves Cardiovascular and Liver Signs of Diet-Induced Metabolic Syndrome in Rats. Nutrients. 2020 Mar 27;12(4):931. doi: 10.3390/nu12040931. PMID 32230955
- [Background] Zhao R, Shen GX. Impact of anthocyanin component and metabolite of Saskatoon berry on gut microbiome and relationship with fecal short chain fatty acids in diet-induced insulin resistant mice. J Nutr Biochem. 2023 Jan;111:109201. doi: 10.1016/j.jnutbio.2022.109201. Epub 2022 Nov 1. PMID 36332818
- [Background] Zhao R, Xiang B, Dolinsky VW, Xia M, Shen GX. Saskatoon berry powder reduces hepatic steatosis and insulin resistance in high fat-high sucrose diet-induced obese mice. J Nutr Biochem. 2021 Sep;95:108778. doi: 10.1016/j.jnutbio.2021.108778. Epub 2021 May 15. PMID 34004342
- [Background] Zhao R, Huang F, Shen GX. Dose-Responses Relationship in Glucose Lowering and Gut Dysbiosis to Saskatoon Berry Powder Supplementation in High Fat-High Sucrose Diet-Induced Insulin Resistant Mice. Microorganisms. 2021 Jul 21;9(8):1553. doi: 10.3390/microorganisms9081553. PMID 34442633
- [Background] Huang F, Zhao R, Xia M, Shen GX. Impact of Cyanidin-3-Glucoside on Gut Microbiota and Relationship with Metabolism and Inflammation in High Fat-High Sucrose Diet-Induced Insulin Resistant Mice. Microorganisms. 2020 Aug 14;8(8):1238. doi: 10.3390/microorganisms8081238. PMID 32824001
- [Background] Zhao R, Khafipour E, Sepehri S, Huang F, Beta T, Shen GX. Impact of Saskatoon berry powder on insulin resistance and relationship with intestinal microbiota in high fat-high sucrose diet-induced obese mice. J Nutr Biochem. 2019 Jul;69:130-138. doi: 10.1016/j.jnutbio.2019.03.023. Epub 2019 Apr 9. PMID 31078906
- [Background] Zhao R, Xie X, Le K, Li W, Moghadasian MH, Beta T, Shen GX. Endoplasmic reticulum stress in diabetic mouse or glycated LDL-treated endothelial cells: protective effect of Saskatoon berry powder and cyanidin glycans. J Nutr Biochem. 2015 Nov;26(11):1248-53. doi: 10.1016/j.jnutbio.2015.05.015. Epub 2015 Jul 17. PMID 26260864
- [Background] Zhao R, Le K, Li W, Ren S, Moghadasian MH, Beta T, Shen GX. Effects of Saskatoon berry powder on monocyte adhesion to vascular wall of leptin receptor-deficient diabetic mice. J Nutr Biochem. 2014 Aug;25(8):851-7. doi: 10.1016/j.jnutbio.2014.03.016. Epub 2014 Apr 13. PMID 24925752